CLINICAL TRIAL: NCT01312389
Title: A Phase I/II Randomized Clinical Trial of Autologous Oxidized Tumor Cell Lysate Vaccine For Recurrent Ovarian, Fallopian Tube or Primary Peritoneal Cancer
Brief Title: A Clinical Trial of Autologous Oxidized Tumor Cell Lysate Vaccine For Recurrent Ovarian, Fallopian Tube or Primary Peritoneal Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Did not meet criteria laid out in Phase 1 to continue to Phase 2
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 29810
Record Dates: First submitted 2011-03-01; First posted 2011-03-10 (Estimated); Results first posted 2021-11-15 (Actual); Last update posted 2021-11-15 (Actual); Status verified 2021-10

CONDITIONS: Ovarian Cancer; Fallopian Tube Cancer; Primary Peritoneal Cancer
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms | interventions — poly(I).poly(c12,U); Heptavalent Pneumococcal Conjugate Vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Phase 2: Arm A (Experimental): 10 patients will receive vaccine (OC-L, an autologous vaccine comprised of autologous oxidized tumor cell lysate, admixed with Montanide ISA 51 VG) injected by intradermal/subcutaneous injection in both groin regions.
  Interventions: Biological: OC-L/Montanide ISA 51 VG; Biological: Prevnar
- Phase 2: Arm B (Experimental): 10 patients will receive vaccine (OC-L, an autologous vaccine comprised of autologous oxidized tumor cell lysate, admixed with Montanide ISA 51 VG) injected by intradermal/subcutaneous injection in both groin regions, administered in combination with intravenous Ampligen.
  Interventions: Biological: OC-L/Montanide ISA 51 VG; Biological: Ampligen; Biological: Prevnar
- Phase 1 (Experimental): 3 patients will be enrolled receiving the vaccine (tumor lysate/Montanide) plus Ampligen using a 3+3 approach. If no DLTs in the first three subjects, we will move to phase II; if one 1/3 subject develops DLTs, we will enroll 3 additional subjects; if 2/6 subjects develop DLTs, we will discontinue the study. Following completion of run---in phase I (3 or 6 subjects), we will transition to Phase 2.
  Interventions: Biological: OC-L/Montanide ISA 51 VG; Biological: Ampligen; Biological: Prevnar

INTERVENTIONS:
Biological: OC-L/Montanide ISA 51 VG — All subjects will receive OC-L/Montanide ISA 51 VG) on day 0, 14,28,42 and 56 with a +/- 5 day window. The vaccine will be divided in two or more intradermal/subcutaneous injections in the groin areas bilaterally.
Biological: Ampligen — All subjects will receive intravenous Ampligen (200mg given by IV infusion 60 +- minutes) 3 times starting 2-3 days after each vaccine administration. Each of the 3 Ampligen (200 mg) infusions will be separated by 2-3 days.
  Arms: Phase 1; Phase 2: Arm B
Biological: Prevnar — A vaccine against Pneumococcus pneumoniae will be given intramuscularly on Day 0 and 14 as positive control of immune responsiveness.

SUMMARY:
This is a Phase I/II randomized study for subjects with recurrent ovarian, fallopian tube or primary peritoneal cancer to determine the feasibility and safety as well as immunogenicity of OC-L, an autologous vaccine comprised of autologous Oxidized tumor Cell Lysate (OC-L) administered by intradermal/subcutaneous injection in combination with Ampligen (poly-l:poly-C12U), a Toll-like receptor 3 agonist. Study duration is 24 months.

DETAILED DESCRIPTION:
This is a Phase I/II randomized study for subjects with recurrent ovarian, fallopian tube or primary peritoneal cancer to determine the feasibility and safety as well as immunogenicity of OC-L, an autologous vaccine comprised of autologous Oxidized tumor Cell Lysate (OC-L) administered by intradermal/subcutaneous injection in combination with Ampligen (poly-l:poly-C12U), a Toll-like receptor 3 agonist. Study duration is 24 months. This study has two Phases eligible subjects enrolled in Phase 1 will receive the OC-L admixed with Montanide ISA 51 with intravenous Ampligen. Subjects enrolled in Phase II will be randomized to two ARMS. This randomized design will allow for the unbiased evaluation and comparison of immune response among the 2 treatment arms. patients will be randomized (10 per treatment arm) in blocks of size 4 or 6, such that treatment assignment will be balanced after each group of 4 or 6 patients has been randomized. ARM A 10 patients will receive OC-L. Arm b 10 patients will receive OC-L with Ampligen. Following each vaccination, subjects in Phase I and Arm B will be given intravenous Ampligen 3 times starting 2-3 days after each vaccine administration. All subjects will receive vaccine on Day 0, 14, 28, 42 and 56. Subjects will receive Prevnar on day 0 and day 14. Subjects will be treated till exhaustion of OC-L or disease progression whichever occurs first subjects will be contacted every 6 months for up to 5 years and then annually for survival. The OC-L study product is manufactured and quality tested at Cell and Vaccine Production Facility and then released to IDS, where it will be admixed with Montanide ISA 51 VG on day of vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Subject has recurrent ovarian (including low malignant potential), fallopian tube or primary peritoneal cancer and has already received front line platinum based chemotherapy prior to recurrence.
* Subject has had prior secondary cytoreductive surgery yielding tumor for Lysate preparation.
* Lysate must meet release criteria.
* Subject has a current largest tumor nodule that is >1 cm CT or MRI.
* Subject is 18 years of age or older.
* Subject has an ECOG performance status of <1.
* Subject has a life expectancy of >6 months.
* Subject must understand and sign the study specific informed consent.
* Subject may have received chemotherapy or other therapy after harvest of tumor and prior to enrollment but must have recovered from toxicities of prior chemotherapy or other therapy (to grade 2 or less).
* Subject may have received prior investigational therapy (including immune therapy).
* Subject may have received prior hormonal therapy.
* Subject may have received prior radiation therapy but must have completed such therapy prior to enrollment.
* Subject who screen fails can be re-enrolled if the causation of the screen fail has been corrected.

Exclusion Criteria:

* Subject for whom tumor lysate does not meet release criteria.
* Subject has a positive serum Yo antibody
* Subject has a chronic or acute hepatitis C infection.
* Subject has a chronic or acute hepatitis B infection.
* Subject has positive test result at the screening visit for one or more of the following: 1. HTLV-1/2 Antibody, 2. Anti-HIV 1/2 Antibody
* Subject requires or is likely to require more than a two-week course of corticosteroids for intercurrent illness. Subject must complete the course of corticosteroids 2 weeks before screening to meet eligibility.
* Subject has renal insufficiency as defined by a serum creatinine > 2.2 mg/dl. Note: If creatinine is greater than 1.5 x ULN, creatinine clearance must be greater than 50 ml/min.
* Subject with liver failure as defined by a serum total bilirubin > 2.0 and /or serum transaminases > 3X the upper limits of normal.
* Subject has any acute infection that requires specific therapy. Acute therapy must have been completed within seven days prior to study enrollment.
* Subject has a serious, non-healing wound, ulcer, or bone fracture.
* Subject has known allergies to reagents used in this study.
* Subject has organ allograft.
* Subject is receiving medications that might effect immune function. Use of H2 antagonists are prohibited, as are all antihistamines five days before and five days after each injection of study vaccine. However, NSAIDS including COX-2 inhibitors, acetaminophen or aspirin are permitted.
* Subject has clinical symptoms or signs of partial or complete gastrointestinal obstruction or requires parenteral hydration and/or nutrition.
* Subject has hematopoietic failure at baseline as defined by one of the following:

  1. Platelets<100,000/mm 3
  2. WBC < 2,500/mm3
  3. Absolute Neutrophil Count (ANC) < 1,500/mm3
  4. Absolute lymphocyte count <200/mm 3
  5. Hematocrit < 30%

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2011-04 (Actual); Primary Completion 2012-05 (Actual); Study Completion 2012-08-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janos Tanyi, MD, Ph.D, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Phase 1 patients were not to continue into Phase 2. If the study had continued, new patients would have been recruited into Phase 2.
Groups:
- Phase 2, Arm A: 10 patients will receive vaccine (OC-L, an autologous vaccine comprised of autologous oxidized tumor cell lysate, admixed with Montanide ISA 51 VG) injected by intradermal/subcutaneous injection in both groin regions.
  OC-L/Montanide ISA 51 VG: All subjects will receive OC-L/Montanide ISA 51 VG) on day 0, 14,28,42 and 56 with a +/- 5 day window. The vaccine will be divided in two or more intradermal/subcutaneous injections in the groin areas bilaterally.
  Ampligen: All subjects will receive intravenous Ampligen (200mg given by IV infusion 60 +- minutes) 3 times starting 2-3 days after each vaccine administration. Each of the 3 Ampligen (200 mg) infusions will be separated by 2-3 days.
  Prevnar: A vaccine against Pneumococcus pneumoniae will be given intramuscularly on Day 0 and 14 as positive control of immune responsiveness.
- Phase 2, Arm B: 10 patients will receive vaccine (OC-L, an autologous vaccine comprised of autologous oxidized tumor cell lysate, admixed with Montanide ISA 51 VG) injected by intradermal/subcutaneous injection in both groin regions, administered in combination with intravenous Ampligen.
  OC-L/Montanide ISA 51 VG: All subjects will receive OC-L/Montanide ISA 51 VG) on day 0, 14,28,42 and 56 with a +/- 5 day window. The vaccine will be divided in two or more intradermal/subcutaneous injections in the groin areas bilaterally.
  Ampligen: All subjects will receive intravenous Ampligen (200mg given by IV infusion 60 +- minutes) 3 times starting 2-3 days after each vaccine administration. Each of the 3 Ampligen (200 mg) infusions will be separated by 2-3 days.
  Prevnar: A vaccine against Pneumococcus pneumoniae will be given intramuscularly on Day 0 and 14 as positive control of immune responsiveness.
Period: Phase 1
Arm/Group | Phase 1 | Phase 2, Arm A | Phase 2, Arm B
Started | 3 | 0 | 0
Completed | 3 | 0 | 0
Not Completed | 0 | 0 | 0
Period: Phase 2
Arm/Group | Phase 1 | Phase 2, Arm A | Phase 2, Arm B
Started | 0 | 0 | 0
Completed | 0 | 0 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: No subjects were enrolled in Phase 2 (Arm A or B)
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1 | Phase 2, Arm A | Phase 2, Arm B | Total
Number analyzed (Participants) | 3 | 0 | 0 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 |  |  | 0
  Between 18 and 65 years | 1 |  |  | 1
  >=65 years | 2 |  |  | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 |  |  | 3
  Male | 0 |  |  | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: Safety will be established by grading the observed toxicities using the NCI Common Toxicity Criteria (CTC Version 4.0). All toxicities observed within 30 days of last vaccination will be included. All patients that receive at least one vaccination will be included in the toxicity analysis.
Time Frame: within 30 days of last vaccination
Population: The study was terminated after the first 3 patients were enrolled in Phase 1
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1 | Phase 2, Arm A | Phase 2, Arm B
Number analyzed (Participants) | 3 | 0 | 0
Participants | 3 |  |

2. Secondary Outcome: Immune Response
Description: Immune response will be evaluated by IFN-g ELISPOT analysis of tumor-reactive T cells, and in HLA-A2+ subjects, by tetramer analysis of Her-2 specific T cells in peripheral blood. Response is defined by a > 3 fold increase relative to pre-vaccination.
Time Frame: within 30 days of vaccination
Population: The study was terminated and the PI has left the institution. Despite all possible efforts to contact the PI/study team members, no data available to be reported.
Arm/Group | Phase 1 | Phase 2, Arm A | Phase 2, Arm B
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: Clinical Response
Description: Clinical Response will be estimated using immune related response criteria ir(RC)
Time Frame: within 30 days of vaccination
Population: as for outcome 2
Arm/Group | Phase 1 | Phase 2, Arm A | Phase 2, Arm B
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 70 days
Description: As there were no participants in Phase 2, there were no participants at risk for any Adverse Events.
Arm/Group | Phase 1 | Phase 2, Arm A | Phase 2, Arm B
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 3/3 | 0/0 | 0/0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1 (N=3) | Phase 2, Arm A (N=0) | Phase 2, Arm B (N=0)
Injection site reaction (Skin and subcutaneous tissue disorders) | 3 (60) | NA | NA
Fatigue (General disorders) | 1 (1) | NA | NA
Flu-like symptoms (General disorders) | 1 (2) | NA | NA
Neuropathy (Nervous system disorders) | 1 (1) | NA | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes